CLINICAL TRIAL: NCT00906386
Title: An Examination of the Efficacy, Safety, and Gender Differences in Using Varenicline as an Aid to Smoking Cessation in a Population of Methadone Maintained Opioid Dependent Patients (Pilot Trial)
Brief Title: Methadone Maintenance Treatment and Smoking Cessation
Acronym: MMTASC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Vancouver Coastal Health (Other Government)
Collaborators: British Columbia Centre of Excellence for Women's Health (Unknown)
Responsible Party: Dr. Milan Khara, Clinical Director, Tobacco Dependence Clinic, Tobacco Dependence Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 60409
Record Dates: First submitted 2009-05-15; First posted 2009-05-21 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2009-05

CONDITIONS: Smoking
Keywords: Varenicline
MeSH Terms: conditions — Smoking | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Varenicline
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Varenicline — oral, 1 mg twice daily, 12 weeks
  Other Names: Champix, Chantix
  Arms: 1
Drug: placebo — oral, 1 mg twice daily, 12 weeks
  Arms: placebo

SUMMARY:
The main hypotheses guiding the study are:

1. Stable methadone maintenance patients receiving varenicline will be more likely to maintain abstinence than patients receiving placebo
2. There will be no differences in the type and number of symptoms reported between stable methadone maintenance patients receiving varenicline and placebo
3. There will be no changes in methadone dosage between abstinent and non-abstinent smokers
4. There will be no differences in efficacy, withdrawal symptoms, and safety of varenicline between male and female participants

DETAILED DESCRIPTION:
1. PURPOSE: The purpose of this placebo controlled study is to determine the efficacy, safety, and gender differences in using varenicline for smoking cessation in a population of stable methadone maintenance patients being treated for Opioid Dependence.
2. HYPOTHESIS:

1.Stable methadone maintenance patients receiving varenicline will be more likely to maintain abstinence than patients receiving placebo 2.There will be no differences in the type and number of symptoms reported between stable methadone maintenance patients receiving varenicline and placebo 3.There will be no changes in methadone dosage between abstinent and non-abstinent smokers 4.There will be no differences in efficacy, withdrawal symptoms, and safety of varenicline between male and female participants

3. JUSTIFICATION: Patients on methadone maintenance treatment have smoking prevalence rates of up 80-90% and consequently disproportionately high mortality compared to the general population. A majority of these patients express a desire to quit but are generally more heavily dependent on nicotine. Randomized controlled trials in non-drug using populations have shown varenicline to be more efficacious for smoking cessation than placebo and other smoking cessation medications. This placebo controlled research protocol will examine varenicline's effect on smoking cessation/reduction and potential sex and gender differences in a population of methadone maintained patients.

4. OBJECTIVES:

Primary outcome:

* Continuous abstinence from smoking during the last 4 weeks of treatment (weeks 9-12).

Secondary outcomes:

* 7-day point prevalence of abstinence
* Continuous abstinence Weeks 9-26
* Sex and gender differences
* Psychological assessment (Beck Depression Inventory)
* Adverse effects (Nausea, Dry mouth, Flatulence, Constipation, Insomnia, -Abnormal dreams, Irritability, Sleep disorder, Headaches, Dizziness e.t.c.)

  5. RESEARCH METHOD: This pilot randomized, double-blind, placebo-controlled trial will be conducted at Vancouver Coastal Health Tobacco Dependence Clinic Vancouver, BC with a 12-week treatment period and follow-up of smoking status to week 26. The intervention will include the use of Varenicline titrated to 1 mg twice daily or placebo for 12 weeks, plus weekly brief smoking cessation counseling.

  6. All significance tests will be 2-tailed with an overall level of significance of a = 0.05. The primary outcome will be the analysis of continuous abstinence using a logistic regression model. The secondary outcomes will be:
  1. the analysis of 7-day abstinence and 9-26 week continuous abstinence using logistic regression analysis.
  2. Minnesota Nicotine Withdrawal Scale, Beck's Depression Inventory, and changes in methadone dose outcome using repeated measures analysis, and
  3. Chi-square tests and t-tests (or Mann-Whitney U) to determine sex and gender differences (male vs female) as well as differences in adverse effects of treatment (varenicline vs placebo)

ELIGIBILITY:
Inclusion Criteria:

* Stable on methadone maintenance (an individual is considered 'stable' if they have had a 4 week constant/fixed dose of methadone by self report and verified by B.C. Pharmanet review)
* Subjects must have smoked at least 10 cigarettes per day during the past year and over the month prior to the screening visit, with no period of abstinence greater than 3 months in the past year
* Ages 19 to 75 years (inclusive) and motivated to quit smoking
* Should read and understand English
* For female subjects:

  * instructed and agrees to avoid pregnancy through 30 days after the last dose of study medication
  * has a negative urine pregnancy test at screening
  * agrees to use birth control method(s) for duration of the study
* Should be available by telephone

Exclusion Criteria:

* Subjects who have used varenicline previously or are currently on other Nicotine Replacement Therapy or pharmacotherapy for smoking cessation (e.g., nicotine patch, zyban or wellbutrin)
* Subjects who have a prior or current history of depression, bipolar affective disorder or a prior or current history of psychotic episodes or suicidal ideation (on the basis of self-report augmented by medical chart review where appropriate and/or corroborating history with previous or current health care provider)
* Subjects who have not reached a stable dose of methadone in their methadone maintenance therapy (4 weeks at a constant/fixed dose of methadone by self-report and verified by B.C. Pharmanet review)
* Pregnancy or currently nursing

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-10 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
7-day point prevalence of abstinence, 9-12 week continuous abstinence, 9-26 week continuous abstinence | 9-12 weeks; 9-26

SECONDARY OUTCOMES:
Sex differences in the efficacy, withdrawal symptoms, and safety of varenicline | week 26

CONTACTS AND LOCATIONS:
Locations (1):
- Three Bridges Community Health Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273